CLINICAL TRIAL: NCT05396950
Title: A Non Randomised Comparative Phase II Trial to Determine the Benefit of Continuous Positive Airway Pressure-assisted Radiotherapy vs Deep Inspiration Breath Hold in Breast Cancer and in Lung & Liver Stereotactic Ablative Body Radiotherapy
Brief Title: CPAP for Motion Management in Breast Radiotherapy; and Lung & Liver SABR
Acronym: CPAP-RT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Waikato Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTN: U1111-1278-1680
Record Dates: First submitted 2022-04-10; First posted 2022-05-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: SABR; CPAP; Breast; Lung; Liver
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Within subject comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP Planned (Experimental): Radiotherapy planning with CPAP in addition to standard plans
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP in conjunction with radiotherapy

SUMMARY:
A phase II trial to determine the proportion of patients where the use of continuous positive airway pressure (CPAP) results in a superior radiation plan compared to standard planning procedures. The rationale for using CPAP with radiotherapy is based on its ability to increase the tidal volume, flatten the diaphragm thus reducing respiratory excursions.The resultant lung hyperinflation and reduced respiratory excursions can be harnessed for radiotherapy purposes by:

1. Displacing the heart away from the radiotherapy field
2. Reducing the volume of functional lung irradiated
3. Reducing the radiotherapy target motion

CPAP has been shown to be superior to free breathing radiotherapy (RT), however it remains unclear how much benefit it confers vs other motion management adjuncts such as deep inspiration breath hold (DIBH) or 4-DCT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine the proportion of patients where the use of CPAP results in a superior radiation plan compared to standard planning procedures in each patient cohort

SECONDARY OBJECTIVES

To determine:

* Impact of CPAP on treatment delivery time;
* Impact of CPAP on total lung volume;
* CPAP compliance;
* Patient experience;

Breast-specific:

• Comparison of organ at risk (OAR) dose constraints between CPAP and deep DIBH)

SABR-specific:

* Internal target volume (ITV) reduction;
* OAR dose constraints between CPAP and standard planning procedures.

Breast cancer patients will undergo normal free breathing and DIBH radiotherapy planning scans. An additional scan with CPAP will be done for the purpose of the study. Radiotherapy plans will be produced on both the DIBH and CPAP planning scans. The planning scan with the best dosimetry will be chosen for treatment. If CPAP has a better radiation plan, then the patient will have CPAP administered during their daily RT. The DIBH plans for each patient, will serve as controls SABR patients will undergo the standard 4-D or breath hold CT and then CPAP CT for the purpose of the study. Respiratory movements will be monitored by Varian RPM system. Radiotherapy plans will be produced from the standard CT and the CPAP CT for comparison.

Patients will be treated on the best plan The trial aim to recruit 70 patients with invasive carcinoma of the breast undergoing adjuvant radiotherapy that includes breast/chest-wall plus regional lymph nodes, and a convenient sample size of those undergoing SABR to lung or liver

ELIGIBILITY:
Inclusion Criteria:

* Any patient with pathologically-confirmed invasive breast cancer and planned for adjuvant radiotherapy to the breast or chest-wall with regional lymph node coverage
* Any patient deemed suitable for lung or liver SABR as per departmental guidelines
* Must have signed written informed consent

Exclusion Criteria:

* Cannot tolerate CPAP e.g due to severe claustrophobia
* Re-irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Radiotherapy Plan Selection | 6-12 months
  To determine the proportion of patients where the use of continuous positive airway pressure (CPAP) results in a superior radiation plan compared to standard planning procedures in each patient cohort

SECONDARY OUTCOMES:
Organ at Risk Dose Constraints | 6-12 months
  Comparison of organ at risk dose constraints between CPAP assisted and standard RT plans
  Breast-specific:
  * A comparison of OAR dose constraints in CPAP vs DIBH including:
    * Mean Heart Dose, V20Gy heart
    * Ipsilateral lung V16Gy and V5Gy SABR-Specific
  * A comparison of OAR dose constraints in CPAP vs DIBH including:
    * Lung V20Gy, Mean Lung Dose
    * Heart V40Gy, Mean heart Dose
    * Liver V15Gy, Mean liver Dose, Liver -GTV
Compliance and Tolerability | 6-12 months
  Assessment of compliance with CPAP as well as documentation of patient experiences
  • Patient experience as documented on a questionnaire after planning CT and on the last week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kenanao D Rantshilane, MBBS, Principal Investigator — Waikato Hospital

IPD SHARING:
Plan to Share IPD: No